CLINICAL TRIAL: NCT06179680
Title: Quantification of White Matter Hyperintensities in Subjects With Amnestic Mild Cognitive Impairment or Alzheimer's Disease
Brief Title: White Matter Hyperintensities in Amnestic Mild Cognitive Impairment or Alzheimer's Disease
Status: Recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Francesco Sardanelli, Prof., IRCCS Policlinico S. Donato
Other Study IDs: WMH-AD
Record Dates: First submitted 2023-11-23; First posted 2023-12-22 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Alzheimer's Disease Group: Description: Individuals diagnosed with Alzheimer's disease. Inclusion Criteria: Participants meeting established criteria for Alzheimer's disease diagnosis, which may include cognitive and memory deficits along with functional impairment.
  Exclusion Criteria: Exclusion of participants with significant comorbidities that could affect cognitive function and those with other forms of dementia.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Amnestic Mild Cognitive Impairment (aMCI) Group: Description: Individuals diagnosed with amnestic mild cognitive impairment. Inclusion Criteria: Participants displaying cognitive decline beyond what is expected for their age but not meeting criteria for a diagnosis of Alzheimer's disease.
  Exclusion Criteria: Exclusion of participants with other neurological conditions that might mimic or contribute to cognitive impairment.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging
- Control Group (Healthy Controls): Description: Individuals without cognitive impairment or neurological disorders.
  Inclusion Criteria: Participants with normal cognitive function for their age, absence of memory complaints, and no history of neurological or psychiatric disorders.
  Exclusion Criteria: Exclusion of individuals with any cognitive impairment, psychiatric disorders, or significant medical conditions affecting cognition.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — MRI Protocol: Uses advanced MRI sequences to examine brain structures and detect white matter issues.
  WMH Assessment: Evaluates white matter health using various methods, including manual and automated tools.
  Neuropsychological Testing: Subjects undergo comprehensive cognitive testing administered by IRCCS Policlinico San Donato's Clinical Psychology Service.
  Follow-up: Patients are monitored for cognitive changes semiannually, with additional assessments for those showing signs of progression. After two years, all patients undergo examination and tests to assess their condition.

SUMMARY:
This study focuses on assessing and measuring white matter hyperintensities in individuals with amnestic mild cognitive impairment (aMCI) or Alzheimer's disease.

Objective:

The primary objective of the study is to quantify the extent and distribution of white matter hyperintensities in the brains of individuals diagnosed with amnestic mild cognitive impairment or Alzheimer's disease. White matter hyperintensities are areas of increased signal intensity observed on brain magnetic resonance imaging (MRI) scans, often associated with various cognitive disorders.

Importance:

Understanding the presence and severity of white matter hyperintensities in individuals with aMCI or Alzheimer's disease is crucial for several reasons. These abnormalities may serve as potential biomarkers, aiding in the early diagnosis and prognosis of cognitive disorders. Additionally, quantifying white matter hyperintensities could contribute to a better comprehension of the underlying neuropathological processes associated with these conditions.

Methods:

The study employs advanced imaging techniques, likely including MRI, to capture and analyze white matter hyperintensities in the brains of participants with amnestic mild cognitive impairment or Alzheimer's disease. The quantification process involves precise measurement and mapping of these hyperintense regions.

Participants:

The study involves individuals diagnosed with amnestic mild cognitive impairment or Alzheimer's disease. Participants will undergo neurological assessments and imaging procedures to facilitate the accurate measurement of white matter hyperintensities.

Expected outcomes:

Researchers anticipate that the quantification of white matter hyperintensities will provide valuable insights into the progression of cognitive disorders. The results may contribute to the development of more targeted and effective diagnostic and therapeutic interventions for individuals with amnestic mild cognitive impairment or Alzheimer's disease.

Conclusion:

This study represents a significant step toward enhancing our understanding of the neuropathological changes associated with amnestic mild cognitive impairment and Alzheimer's disease. By focusing on the quantification of white matter hyperintensities, researchers aim to uncover potential markers for early detection and monitoring of these cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with amnestic Mild Cognitive Impairment (aMCI) or Alzheimer's Disease (AD) based on clinical assessments.
* Individuals undergoing brain magnetic resonance imaging (MRI) at the IRCCS Policlinico San Donato as part of routine diagnostic procedures.
* Age-matched and gender-matched healthy control subjects for comparison.

Exclusion Criteria:

* Individuals with cognitive impairment other than amnestic MCI or AD.
* History of significant neurological disorders (other than MCI or AD) that may impact the study outcomes.
* Presence of contraindications for undergoing MRI procedures.
* Any serious medical or psychiatric condition that, in the judgment of the researchers, may interfere with the study participation or compromise the validity of the results.
* Known history of alcohol or substance abuse that may affect cognitive function.
* Inability or unwillingness to provide informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients with amnestic Mild Cognitive Impairment (aMCI):
  These individuals have been clinically diagnosed with aMCI, a condition characterized by noticeable memory impairment beyond what is expected for age but not meeting the criteria for a diagnosis of Alzheimer's Disease.
  Patients with Alzheimer's Disease (AD):
  Participants diagnosed with Alzheimer's Disease based on clinical assessments.
  Healthy Control Subjects:
  Age-matched and gender-matched individuals without cognitive impairment or significant neurological disorders.
Sampling Method: Non-Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
White Matter Hyperintensity burden | 24 months
  The primary objective is to study the difference in terms of White Matter Hyperintensity (WMH) burden normalized for intracranial volume (primary outcome) between patients with Alzheimer's Disease (AD) and control subjects. This forms the basis for calculating the sample size for prospective recruitment.

SECONDARY OUTCOMES:
Spatial distribution pattern | 24 months
  Evaluate the potential relationship between the extent of WMH burden, both total and specifically their spatial distribution pattern, and the risk of progression to AD dementia in patients with amnestic Mild Cognitive Impairment (aMCI).
TRACE4AD classifier | 24 months
  Assess whether the WMH burden, in conjunction with voxel-based and volumetric analysis of gray matter and neuropsychological test results, can contribute to predicting the progression of aMCI to AD, as defined by the TRACE4AD classifier.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milano, Italy

IPD SHARING:
Plan to Share IPD: No